CLINICAL TRIAL: NCT02192333
Title: Young Adult Cancer Survivor Network Study of the Essential Elements of Care (YA-EEC-14)
Brief Title: Survivorship Care in Reducing Symptoms in Young Adult Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Livestrong Foundation (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 9161; NCI-2014-01325 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9161 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG1001123 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2014-07-15; First posted 2014-07-16 (Estimated); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Breast Carcinoma; Cancer Survivor; Depression; Fatigue; Leukemia; Lymphoma; Malignant Bone Neoplasm; Malignant Digestive System Neoplasm; Malignant Female Reproductive System Neoplasm; Malignant Male Reproductive System Neoplasm; Pain; Sleep Disorder; Soft Tissue Sarcoma
MeSH Terms: conditions — Breast Neoplasms; Depression; Fatigue; Leukemia; Lymphoma; Bone Neoplasms; Gastrointestinal Neoplasms; Pain; Sleep Wake Disorders; Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (usual care) (No Intervention): Participants receive usual care. After 12 months, participants may receive a survivorship clinic visit and boosters as in Arm II.
- Arm II (survivorship care) (Experimental): Participants attend a survivorship clinic visit that includes care plans, screening recommendations, physician coordination, health promotion education, symptom management and palliative care, late effects education, psychosocial and medical assessments, and referrals for services and care as appropriate. Participants also receive phone-based survivorship boosters over approximately 15-30 minutes at 4-8 weeks and 12-16 weeks after the initial clinic visit.
  Interventions: Procedure: Management of Therapy Complications; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Behavioral: Telephone-Based Intervention

INTERVENTIONS:
Procedure: Management of Therapy Complications — Receive survivorship care
  Arms: Arm II (survivorship care)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
  Arms: Arm II (survivorship care)
Other: Questionnaire Administration — Ancillary studies
  Arms: Arm II (survivorship care)
Behavioral: Telephone-Based Intervention — Receive phone-based booster intervention
  Arms: Arm II (survivorship care)

SUMMARY:
This randomized clinical trial studies survivorship care in reducing symptoms in young adult cancer survivors. Survivorship care programs that identify the needs of young adult cancer survivors and ways to support them through the years after treatment may help reduce symptoms, such as pain, fatigue, sleep disturbance, depression, and distress, in young adult cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test the impact of providing the essential elements of survivorship care on survivorship outcomes as indicated by reduction in symptoms (pain, fatigue, sleep disturbance, depression, distress) in young adult cancer survivors diagnosed with cancer between the ages of 18 and 39 years when compared with usual care.

SECONDARY OBJECTIVES:

I. To improve confidence in survivorship knowledge and promote healthy lifestyle behaviors.

II. To provide evidence on barriers, needs and care preferences that will support long term follow-up recommendations for this population.

OUTLINE: Participants categorized as high-need are randomized to 1 of 2 arms. Participants categorized as low-need are assigned to Arm I.

ARM I: Participants receive usual care. After 12 months, participants may receive a survivorship clinic visit and boosters as in Arm II.

ARM II: Participants attend a survivorship clinic visit that includes care plans, screening recommendations, physician coordination, health promotion education, symptom management and palliative care, late effects education, psychosocial and medical assessments, and referrals for services and care as appropriate. Participants also receive phone-based survivorship boosters over approximately 15-30 minutes at 4-8 weeks and 12-16 weeks after the initial clinic visit.

After completion of study, participants are followed up at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled on phase 1 of the study are eligible (and/or if recruited from tumor registry or clinic follow-up schedules)
* Diagnosed with invasive malignancy including: breast, gastrointestinal track, female or male genitourinary system, sarcoma of bone or soft-tissue, leukemia and lymphoma
* Treated at one of the Survivorship Centers of Excellence or their community affiliates
* Received a therapeutic intervention with at least one of the following modalities: surgery, cytotoxic chemotherapy, biological or targeted agents, radiation therapy (any modality)
* Currently between 1.0 and 4.99 years from the completion of active cancer-directed therapy (cytotoxic chemotherapy, radiation therapy and/or definitive surgical intervention)
* Patient must still be in active follow-up: seen for a follow-up visit in the participating center at least once in the 3 years prior to enrollment and/or scheduled to be seen for follow-up in the next 6 months (i.e. in active follow-up)
* May be receiving "maintenance" therapy that has a goal of prevention of recurrence but there should be no expectations for further active treatment
* Able to read and speak English adequate to complete the patient-reported outcomes (PRO) assessment

Exclusion Criteria:

* Prior visit to a survivorship clinic or previously provided with a treatment summary and care plan

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 390 (Actual)
Dates: Start 2015-08-03 (Actual); Primary Completion 2017-10-07 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Mean of the two z scores of the two highest scores for the symptoms that determined the participant's eligibility as "high need" assessed using patient-reported outcomes (PRO) survey | At 6 months
  Mean scores for the primary outcome measures will be compared between the study using standard methods. Two-sided significance levels will be set at an alpha level of 0.05.

SECONDARY OUTCOMES:
Barriers to health care assessed using the patient-reported outcomes (PRO) survey | Up to 12 months
  Will be examined in an exploratory manner, utilizing similar methods as those described for the primary endpoints for dichotomized versions of the outcomes, using standard cutoff values, where available.
Change in depression assessed using the patient-reported outcomes (PRO) survey | Baseline to up to 12 months
  Will be examined in an exploratory manner, utilizing similar methods as those described for the primary endpoints for dichotomized versions of the outcomes, using standard cutoff values, where available. The mean differences in other continuous valued outcomes will be evaluated using standard t-tests or linear regression models, as appropriate.
Change in distress assessed using the patient-reported outcomes (PRO) survey | Baseline to up to 12 months
  Will be examined in an exploratory manner, utilizing similar methods as those described for the primary endpoints for dichotomized versions of the outcomes, using standard cutoff values, where available. The mean differences in other continuous valued outcomes will be evaluated using standard t-tests or linear regression models, as appropriate.
Change in fatigue assessed using the patient-reported outcomes (PRO) survey | Baseline to up to 12 months
  Will be examined in an exploratory manner, utilizing similar methods as those described for the primary endpoints for dichotomized versions of the outcomes, using standard cutoff values, where available. The mean differences in other continuous valued outcomes will be evaluated using standard t-tests or linear regression models, as appropriate.
Change in pain assessed using the patient-reported outcomes (PRO) survey | Baseline to up to 12 months
  Will be examined in an exploratory manner, utilizing similar methods as those described for the primary endpoints for dichotomized versions of the outcomes, using standard cutoff values, where available. The mean differences in other continuous valued outcomes will be evaluated using standard t-tests or linear regression models, as appropriate.
Change in sleep assessed using the patient-reported outcomes (PRO) survey | Baseline to up to 12 months
  Will be examined in an exploratory manner, utilizing similar methods as those described for the primary endpoints for dichotomized versions of the outcomes, using standard cutoff values, where available. The mean differences in other continuous valued outcomes will be evaluated using standard t-tests or linear regression models, as appropriate.
Confidence in survivorship information assessed using the patient-reported outcomes (PRO) survey | Up to 12 months
  Will be examined in an exploratory manner, utilizing similar methods as those described for the primary endpoints for dichotomized versions of the outcomes, using standard cutoff values, where available.
General health assessed using the patient-reported outcomes (PRO) survey | Up to 12 months
  Will be examined in an exploratory manner, utilizing similar methods as those described for the primary endpoints for dichotomized versions of the outcomes, using standard cutoff values, where available.
Health behaviors assessed using the patient-reported outcomes (PRO) survey | Up to 12 months
  Will be examined in an exploratory manner, utilizing similar methods as those described for the primary endpoints for dichotomized versions of the outcomes, using standard cutoff values, where available.
Health care utilization assessed using the patient-reported outcomes (PRO) survey | Up to 12 months
  Will be examined in an exploratory manner, utilizing similar methods as those described for the primary endpoints for dichotomized versions of the outcomes, using standard cutoff values, where available.
Medications assessed using the patient-reported outcomes (PRO) survey | Up to 12 months
  Will be examined in an exploratory manner, utilizing similar methods as those described for the primary endpoints for dichotomized versions of the outcomes, using standard cutoff values, where available.
Mood and worries assessed using the patient-reported outcomes (PRO) survey | Up to 12 months
  Will be examined in an exploratory manner, utilizing similar methods as those described for the primary endpoints for dichotomized versions of the outcomes, using standard cutoff values, where available.
Musculoskeletal symptoms assessed using the patient-reported outcomes (PRO) survey | Up to 12 months
  Will be examined in an exploratory manner, utilizing similar methods as those described for the primary endpoints for dichotomized versions of the outcomes, using standard cutoff values, where available.
Neuropathy assessed using the patient-reported outcomes (PRO) survey | Up to 12 months
  Will be examined in an exploratory manner, utilizing similar methods as those described for the primary endpoints for dichotomized versions of the outcomes, using standard cutoff values, where available.
Post-traumatic stress assessed using the patient-reported outcomes (PRO) survey | Up to 12 months
  Will be examined in an exploratory manner, utilizing similar methods as those described for the primary endpoints for dichotomized versions of the outcomes, using standard cutoff values, where available.
Quality of life assessed using the patient-reported outcomes (PRO) survey | Up to 12 months
  Will be examined in an exploratory manner, utilizing similar methods as those described for the primary endpoints for dichotomized versions of the outcomes, using standard cutoff values, where available.
Reclassification of subject from high need to low need | At 6 months
  Reclassification of subject from high need to low need is defined as the high need subject no longer has scores above the cut-off level on 2 or more symptoms scales (depression, distress, insomnia, fatigue, pain) assessed using the PRO survey. The 5 symptom scales are categorized based on the following cut points to define "high need": pain score >= 5, fatigue score >= 3, insomnia score of no insomnia, distress score > 1.1, and depression score >= 10.
Reproductive health assessed using the patient-reported outcomes (PRO) survey | Up to 12 months
  Will be examined in an exploratory manner, utilizing similar methods as those described for the primary endpoints for dichotomized versions of the outcomes, using standard cutoff values, where available.
Sexual function assessed using the patient-reported outcomes (PRO) survey | Up to 12 months
  Will be examined in an exploratory manner, utilizing similar methods as those described for the primary endpoints for dichotomized versions of the outcomes, using standard cutoff values, where available.
Social support assessed using the patient-reported outcomes (PRO) survey | Up to 12 months
  Will be examined in an exploratory manner, utilizing similar methods as those described for the primary endpoints for dichotomized versions of the outcomes, using standard cutoff values, where available.

CONTACTS AND LOCATIONS:
Overall Officials: K. Scott Baker, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (6):
- United States (6):
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

REFERENCES:
- [Derived] Hall AG, Syrjala KL, Ketterl TG, Ganz PA, Jacobs LA, Palmer SC, Partridge A, Rajotte EJ, Mueller BA, Baker KS. Socioeconomic Factors and Adherence to Health Care Recommendations in Adolescent and Young Adult Cancer Survivors. J Adolesc Young Adult Oncol. 2023 Oct;12(5):701-709. doi: 10.1089/jayao.2022.0109. Epub 2023 Feb 13. PMID 36779982
- [Derived] Syrjala KL, Walsh CA, Yi JC, Leisenring WM, Rajotte EJ, Voutsinas J, Ganz PA, Jacobs LA, Palmer SC, Partridge A, Baker KS. Cancer survivorship care for young adults: a risk-stratified, multicenter randomized controlled trial to improve symptoms. J Cancer Surviv. 2022 Oct;16(5):1149-1164. doi: 10.1007/s11764-021-01105-8. Epub 2021 Sep 29. PMID 34590205